CLINICAL TRIAL: NCT04393792
Title: Can a Sinus Rinse and Mouth Wash Reduce Viral Load in COVID-19 Positive Individuals and Their Co-residents?
Brief Title: SINUS WASH Pilot Study in Adults Testing Positive for COVID-19
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hampshire Hospitals NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SPON-AK-0420; 2020-001721-31 (EudraCT Number)
Record Dates: First submitted 2020-05-18; First posted 2020-05-19 (Actual); Last update posted 2021-09-17 (Actual); Status verified 2021-09

CONDITIONS: Coronavirus Infection
Keywords: COVID-19; sinus rinse; mouth wash; povidone-iodine; coronavirus; Wuhan
MeSH Terms: conditions — Coronavirus Infections; COVID-19 | interventions — Povidone-Iodine; Saline Solution

STUDY DESIGN:
Intervention Model Description: unblinded parallel group design with 1:1 randomised allocation to treatment or control
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Povidone-Iodine (Active Comparator): 0.23% sinus rinse and mouthwash three times daily (tds) for days 1-3 of study
  Interventions: Drug: Povidone-Iodine
- Normal Saline (Placebo Comparator): sinus rinse and mouthwash three times daily (tds) for days 1-3 of study
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: Povidone-Iodine — 0.23% three times daily (tds) for 3 days
  Other Names: Videne Antiseptic Solution
  Arms: Povidone-Iodine
Drug: Normal saline — 0.9% three times daily (tds) for 3 days
  Arms: Normal Saline

SUMMARY:
COVID-19 is highly infectious and transmission of the virus is thought to be similar to that of influenza which can be transferred through droplets released when a person coughs, sneezes or talks. Studies have shown that nasal rinsing and mouth washes may be an important way to deliver treatments that could reduce the amount of a virus that is present in the nose and mouth. This also could mean that there is less virus available to pass on to others. We want to see if the use of nose rinses and mouth washes using Povidone-Iodine will reduce the the amount of virus in the nose and throat of people who have tested positive for COVID-19 disease and also reduce the spread of infection within their household.

DETAILED DESCRIPTION:
COVID-19 is highly infectious and transmission of the virus is thought to be similar to that of influenza which can be transferred through droplets released when a person coughs, sneezes or talks. Studies have shown that nasal rinsing and mouth washes may be an important way to deliver treatments that could reduce the amount of a virus that reaches other parts of the body. This also could mean that there is less virus available to pass on to others.

We want to see if the use of nasal rinsing and mouth washes will reduce the spread of infection within your household by reducing and removing the virus from your mouth and nose.

Once the participants have been recruited they will be randomly allocated to one of two groups. Each arm will have the same number of participants. The two arms will be :

1. nose rinse and mouthwash with Isotonic saline alone. This will be the control arm.
2. nose rinse and mouthwash with Povidone-Iodine taken 3 times a days for three days.

Before treatment begins, each participant will have one pre-treatment swab of the back of the nose and the back of the throat taken.

Once allocated each participant will be asked to have 4 further swabs of the mouth and nose taken on days 2,4,7 & 14.

Participants will be patients and healthcare staff who have tested positive for COVID-19. Healthcare staff who are self isolating will also asked their co-residents/family members at home to take the treatment and provide swabs in the same manner.

Participants who are patients and are admitted to hospital will be well enough to perform the nasal rinses and mouth washes as treatments and provide the same swabs.

All participants will be provided with informational videos on how to do the treatments and how to take the swabs. Participants who are not healthcare staff will have swabs taken as part of the local drive through testing service.

All participants will be asked to download a free smartphone app (Umotif) to upload information about daily symptoms and whether they have provided swabs on the required days.

The swabs will be tested for the amount of virus in the labs at Hampshire Hospitals NHS Foundation Trust and analysed to determine if the treatment arm of Povidone-Iodine is reducing the amount of virus compared to the isotonic saline arm.

All results will be anonymised prior to analysis. The study team will know the participants' study-specific data; no personal data about participants will be used without their explicit consent and only for the purposes of protocol adherence and data to answer the study question.

Once the last swab has been taken and delivered to the laboratory, the trial will have ended for that participant. Results of the swabs will be part of the study data and collated in readiness for analysis by the study statistician.

The results will be made available for peer-reviewed publication and presentation at conferences.

ELIGIBILITY:
Inclusion Criteria:

* Healthcare worker OR patient on a general ward who has had a positive COVID-19 test OR a person who is co-residing with an affected staff member or patient who is now at home in self-isolation.
* capable of giving informed consent
* able to self-administer the sinus rinses and mouth washes
* able to have healthcare professional-led swabs OR self-administer the oral and nasopharyngeal swabs
* aged 18 years and over.

Exclusion Criteria:

* not capable of giving informed consent
* unable to self-administer the sinus rinses and mouth washes
* unable to have healthcare professional-led swabs OR self-administer the oral, nasal and/OR nasopharyngeal swabs
* unable to send swabs to the study team via the approved methods described in participant information leaflet and protocol
* under 18 years of age.
* known hypersensitivity to Iodine
* at risk of aspiration due to an unsafe swallow
* hyperthyroidism or other manifest thyroid diseases
* herpetiform dermatitis (Duhring's disease)
* planned or undergoing radioiodine treatment
* actively Breastfeeding
* pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-05-05 (Actual); Primary Completion 2022-03 (Estimated); Study Completion 2022-03 (Estimated)

PRIMARY OUTCOMES:
Change in viral load in the oral and nasopharyngeal cavity | Day 0, 2, 3, 7, 14
  viral load as measured by real time polymerase chain reaction (PCR)

SECONDARY OUTCOMES:
Symptom severity in primary participants and co-residents | Days 0 to 14
  Visual analogue score 1-5 per symptom via a smartphone app

CONTACTS AND LOCATIONS:
Overall Officials: Afroze Khan, MBBS MRCS, Principal Investigator — Hampshire Hospitals NHS Foundation Trust
Locations (1):
- Hampshire Hospitals NHS Foundation Trust, Basingstoke, Hampshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No